CLINICAL TRIAL: NCT03901638
Title: Gut Microbiota Alteration and Improvement of Ataxia in Patients of Multiple System Atrophy Treating With Tllsh2910 - a Randomized, Placebo-controlled, Double-blinded, Cross-over, Single-center Clinical Trial
Brief Title: Tllsh2910 for Ataxia and Gut Microbiota Alteration in Patients of Multiple System Atrophy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Project replanning
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201810015MINC
Record Dates: First submitted 2019-03-24; First posted 2019-04-03 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2020-04

CONDITIONS: Ataxia, Cerebellar; Multiple System Atrophy
Keywords: multiple system atrophy, cerebellar ataxia, NMDA, microbiota
MeSH Terms: conditions — Cerebellar Ataxia; Multiple System Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tllsh2910 to placebo (Experimental): Tllsh2910 160mg per day for 12 weeks with wash-out period 12 weeks and subsequent placebos for 12 weeks.
  Interventions: Drug: Tllsh2910; Drug: Placebo
- Placebo to Tllsh2910 (Experimental): Placebos for 12 weeks with wash-out period 12 weeks and subsequent Tllsh2910 160mg per day for 12 weeks
  Interventions: Drug: Tllsh2910; Drug: Placebo

INTERVENTIONS:
Drug: Tllsh2910 — Tllsh2910 80mg twice per day orally for 12 weeks
Drug: Placebo — Placebo

SUMMARY:
Multiple system atrophy (MSA) is a fetal, rare neurodegenerative disease presenting with parksinonism, autonomic dysfunction, and cerebellar ataxia. Numerous anti-parkinsonism agents have been developed. However, no medication has yet been proven effective for the symptomatic or even causative treatment in cerebellar ataxia. To our knowledge, cerebellar N-methyl-D- aspartic acid (NMDA) receptors play a special role in the modulation of motor learning and coordination. Tllsh2910, a NMDA modulator, has been found to attenuate the ataxic gait in the mouse model. Here, we designed a large-scale double-blind randomized controlled, cross-over phase III trial to investigate the efficacy of Tllsh2910 in neurodegenerative ataxic patients and the association of gut microbiota change.

DETAILED DESCRIPTION:
The study is terminated prematurely due to project replanning and difficulty in recruitment during the pandemic. The overall sample size is not adequate to meet the requirement of estimated power. The statistical results will be investigated. No severe drug-related adverse events were reported during the study period.

ELIGIBILITY:
Inclusion Criteria:

* 1. Clinically confirmed cerebellar ataxia with a SARA total score ≥ 3 (range 0-40).
* 2. Clinical diagnosis of probable or possible MSA-C.
* 3. Patients older than 18 years old and younger than 80 years old.

Exclusion Criteria:

* 1. Major systemic diseases such as hepatic, renal or heart failure, malignancy, stroke.
* 2. Concomitant medication which inhibit CYP2C19 enzyme such as Clopidogrel, cimetidine, fluconazole, ketoconazole, voriconazole, etravirine, fluoxetine, fluvoxamine, ticlopidine.
* 3. Pregnancy and/or breastfeeding.
* 4. Acute diseases that might interfere with the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
=Scale for the assessment and rating of ataxia (SARA) score | Baseline, 12 weeks, 24 weeks, 36 weeks
  SARA is an 8-item performance based scale with gait, stance, sitting, speech disturbance, finger chase, nose-finger test, fast alternative hand movements, and heel-shin slide, yielding a total score of 0 (no ataxia) to 40 (most severe ataxia). The change in the SARA score will be recorded from period-level baseline to the end of the 12-week, 24-week, 36-week treatment period.

SECONDARY OUTCOMES:
International Cooperative Ataxia Rating Scale (ICARS) score | Baseline, 12 weeks, 24 weeks, 36 weeks
  ICARS is an 19-item performance based scale with 4 subscales of postural and gait disturbances, kinetic function, speech disorders, and oculomotor disorders, yielding a total score of 0 (no ataxia) to 100 (most severe ataxia). The change in the ICARS score will be measured from period-level baseline to the end of the 12-week, 24-week, 36-week treatment period.
Unified multiple system atrophy rating scale (UMSARS) Part II score | Baseline, 12 weeks, 24 weeks, 36 weeks
  UMSARS is an validated 26-items scale for multiple system atrophy with 4 subscales of historical review, motor examination scale, autonomic examination, and global disability scale. The Part II is a performance based subscale, yield a total score of 0 (no motor impairment) to 56 (most severe motor impairment). The change in the UMSARS Part-II score will be measured from period-level baseline to the end of the 12-week, 24-week, 36-week treatment period.
The composition change of gut microbiota | Baseline, 12 weeks
  The gut microbiota will be measured at baseline and 12th weeks.
The change of total time needed for a 8-meter walking test | Baseline, 12 weeks, 24 weeks, 36 weeks
  Total time of 8-meter walking test will be measured from period-level baeline to the end of the 12-week, 24-week, and 36-week.
The change of the World Health Organization Quality of Life (WHOQOL-BREF) scale | Baseline, 12 weeks, 24 weeks, 36 weeks
  The WHOQOL-BREF scale is a 28-item questionnaire about quality of life. The change of WHOQOL-BREF scores will be measured at baseline, 12-week, 24-week, and 36-week.
The total time needed for 9 hole peg test | Baseline, 12 weeks, 24 weeks, 36 weeks
  The total time needed for 9 hole peg test will be measured at the baseline, 12-week, 24-week, and 36-week.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Hwei Tai, Principal Investigator — National Taiwan University Hospital (NTUH)
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No